CLINICAL TRIAL: NCT04597853
Title: Assessment of Lung Mechanics in SARS-CoV-2/ COVID-19 Acute Respiratory Distress Syndrome: A Holistic, Longitudinal Analysis of the Lung-heart-ventilator Interaction
Brief Title: Assessment of Lung Mechanics in COVID-19 Acute Respiratory Distress Syndrome
Acronym: LungMechCoV-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01999
Record Dates: First submitted 2020-10-19; First posted 2020-10-22 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Covid19; ARDS
Keywords: lung mechanics; heart-lung interaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessment of lung mechanics and heart-lung interactions — Impedance tomography, right-heart catheterization, oesophageal pressure measurements, indirect calorimetry and classic mechanical ventilation parameters

SUMMARY:
This study is meant to assess the lung mechanics in SARS-CoV-2 induced acute respiratory failure. A precise characterisation of lung mechanics and heart-lung-interactions might allow a better understanding of SARS-CoV-2 induced acute respiratory failure and thus lead to better mechanical ventilation strategies.

This monocentric, observational study of critically ill COVID-19 patients in the ICU, will employ impedance tomography, right-heart catheterization, oesophageal pressure measurements, indirect calorimetry as well as classic mechanical ventilation parameters to characterise the mechanical characteristics of the lung as well as the heart-lung interactions in SARS-CoV-2 induced acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection
* Moderate to Severe ARDS after Berlin Classification at PEEP 5
* Admission to the Institute of Intensive Care of the University Hospital Zurich
* Invasive Mechanical Ventilation
* Signed Study Informed Consent or emergency procedure according to article 30 HFG

Exclusion Criteria:

* Pregnant or breast feeding patients
* Age <18 years
* Presumed rejection of the study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project population targeted with this research, consists of a critically ill COVID-19 diagnosed population being admitted to the Institute of Intensive Care of the University Hospital Zurich and treated with mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Time dependent compliance change | Mixed Model Assessment of compliance over time until extubation (measurements every 2 days up to 90 days)
  Compliance change over the length of mechanical ventilation
PEEP and time dependent change in dead space | Mixed Model Assessment of Dead Space over time until extubation (measurements every 2 days up to 90 days)
  Change in Dead Space over the length of mechanical ventilation
PEEP and time dependent change in shunt fraction | Mixed Model Assessment of shunt fraction over time until extubation (measurements every 2 days up to 90 days)
  Change in shunt fraction over the length of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Philipp K Buehler, MD, Principal Investigator — Institute of Intensive Care Medicine, University Hospital Zurich
Locations (1):
- Institute of Intensive Care Medicine, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided